CLINICAL TRIAL: NCT03440892
Title: Longitudinal Observational Study on Rheumatoid Arthritis Patients: Effects of Antirheumatic Treatment on Serum Levels of Survivin
Brief Title: Effects of Antirheumatic Treatment on Levels of Survivin in Rheumatoid Arthritis Patients
Acronym: SurviTreat
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: Survivin in Treatment
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis
Keywords: survivin; biomarker of pharmacological response; antirheumatic treatment; methotrexate; sulfasalazin; abatacept; tocilizumab; tofacitinib/baricitinib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Sulfasalazine; Abatacept; tocilizumab; tofacitinib; baricitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: methotrexate; Drug: sulfasalazine; Drug: abatacept; Drug: tocilizumab; Drug: tofacitinib/baricitinib

INTERVENTIONS:
Drug: methotrexate — folate antagonist
Drug: sulfasalazine — Immunomodulatory
  Other Names: Salazopyrin
Drug: abatacept — Targeting CTLA-4 (fusion protein composed of the Fc region of the immunoglobulin IgG1 fused to the extracellular domain of CTLA-4)
  Other Names: Orencia
Drug: tocilizumab — IL-6 receptor antagonist
  Other Names: RoActemra
Drug: tofacitinib/baricitinib — JAK inhibitor
  Other Names: Xeljanz/Olumiant

SUMMARY:
To validate the utility of survivin as a biomarker of pharmacological response to therapeutic intervention in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
In a prospective observational study the investigators aim to study the ability of modern antirheumatic treatments to suppress levels of survivin in sera. Rheumatoid arthritis patients scheduled to start new pharmacological treatment will be followed for a period of 6 months. No intervention or influence on choice of treatment will be performed, the decision of new/other medication is entirely made by the patient and their rheumatologist. The study entails addition of survivin analyse (1 vial of sera) before and after start of new treatment. Data concerning survivin levels, disease activity and other clinical parameters before and after start of new treatment will also be analysed. The patients will leave sera for survivin analyse at baseline and 3 and 6 months after start of new treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the RA classification criteria according to the ACR/EULAR

Exclusion Criteria:

* Patients at stable/unchanged anti-rheumatic treatment
* Other serious physical or mental illness
* Lack of knowledge in Swedish making answering the questionnaires impossible

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Survivin status | 6 months
  Patients with a survivin level of over 0.45 ng/ml are considered to be survivin positive.
  Patients with survivin levels under 0.45 ng/ml are considered to be survivin negative
  A change from survivin positive to survivin negative (or vice versa) equals conversion of survivin status.

SECONDARY OUTCOMES:
Disease activity (DAS28) | 6 months
  Disease activity, DAS28, is calculated using a specific formula based on:
  * number of painful joints from 28 joints
  * number of swollen joints from 28 joints
  * erythrocyte sedimentation rate (ESR) or C reactive protein (CRP)
  * patient's global assessment of disease activity on a 100 mm visual analogue scale (VAS)
  DAS thresholds:
  DAS28 below 3.2: low disease activity DAS28 over 3.2 and under 5.1: moderate disease activity DAS28 above 5.1: high disease activity DAS28 lower than 2.6: remission
Response to treatment | 6 months
  The EULAR response criteria classify patients as good, moderate, or non-responders, using the change in DAS28 and the level of DAS28 reached. A patient must show a significant change as well as low disease activity to be classified as a good responder.
  Good responder: DAS28 scores ≤ 3.2 with reductions in DAS28 >1.2 Moderate responder: DAS28 scores > 3.2 with reductions in DAS28 >1.2 Non-responder: reductions in DAS28 ≤ 0.6

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Rheumatology and Inflammation research, Gothenburg, Sweden